CLINICAL TRIAL: NCT02652572
Title: Open Label Pharmacokinetic Study of Granexin® Gel in Patients With Venous Leg Ulcers
Brief Title: Safety Study to Examine the Systemic Exposure of Granexin® Gel After Topical Application to Venous Leg Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xequel Bio, Inc. (Other)
Collaborators: Spartanburg Regional Healthcare System (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VLU-PK-300
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Venous Leg Ulcer
Keywords: Granexin; venous leg ulcer; pharmacokinetic study; FirstString Research
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Granexin® gel plus standard-of-care (Experimental): Granexin® gel will be applied topically to diabetic foot ulcer(s) on Day 0 (baseline), Day 3, and Day 7. In addition, standard-of-care treatment will be applied to the ulcer(s) at Screening, Day 0, Day 3, and Day 7.
  Interventions: Drug: Granexin

INTERVENTIONS:
Drug: Granexin — Granexin® gel will be dispensed directly from a 5 gram laminate tube and will be spread and smoothed directly over the wound surface in full contact with the wound bed to obtain an even, uniform layer on Day 0 (baseline), Day 3, and Day 7.

SUMMARY:
The purpose of this study is to determine the systemic exposure of Granexin® gel after topical application to human subjects' venous leg ulcers.

DETAILED DESCRIPTION:
The objective of this study is to ascertain the systemic exposure of the active ingredient in Granexin® gel (aCT1 peptide) after topical application to venous leg ulcers using pharmacokinetic analysis. It is planned that a total of 16 patients with venous leg ulcers will receive Granexin® gel treatment plus standard of care in this one arm study. The study includes a screening period (1 week) and a treatment period (1 week) which occur sequentially for a given patient.The baseline day, which demarcates the beginning of the treatment period, is the designated as Day 0. Screening procedures are initially conducted on Day -7.

A target venous leg ulcer is identified at screening and patient eligibility is confirmed at screening and then again at the beginning of the Day 0 (baseline) visit. A patient enrolled in the study may have multiple ulcers on the same or either leg; in this case, all ulcers will be treated with Granexin® gel, but only ulcer(s) meeting the following criteria will be designated as the target ulcer(s) and will determine eligibility: >15cm2 of least 4 weeks duration in post debridement.

The treatment period for a given patient begins on Day 0 and ends one week later; the last scheduled day of the treatment period is designated as Day 7. During each treatment period, each patient is scheduled to receive topical treatment with study drug gel (3 applications total) administered by study staff at scheduled study site visits at each of the following time points: Day 0 , Day 3, and Day 7. All patients, regardless of treatment assignment, also receive standard-of-care treatment at scheduled study visits during the treatment period.

Study drug pre-application blood samples will be collected from each patient at Day 0, Day 3, and Day 7. Study drug post-application blood samples will be collected at Day 0 and Day 7 at time points specified in the protocol. These blood samples will be shipped to a designated laboratory for pharmacokinetic analysis.

Safety will be assessed during the treatment period by monitoring adverse events, measuring vital signs at each visit, performing physical examinations, electrocardiograms (ECG), as well as pharmacokinetic (PK) blood analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosis of venous leg ulcer(s), as clinically determined by the investigator by a positive venous reflux test (venous refilling <20 seconds) using Doppler ultrasound for at least 4 weeks prior to screening day, which have not adequately responded to conventional ulcer therapy.
3. Designated venous leg ulcer meets the following criteria at both the screening and baseline visits. If the patient has multiple ulcers, at least one ulcer must meet the following criteria at both the screening and baseline visits:

   1. Present for at least 4 weeks
   2. CEAP Classification Stage 6
   3. Surface ulcer with an area > 15cm2 post debridement
   4. Viable, granulating wound (investigator discretion)
4. Ulcers that extend through the epidermis but not through the muscle, tendon, or bone (Stage II or III ulcers as defined by the IAET).
5. Female patients of childbearing potential must have a negative pregnancy test at screening and must agree to use hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence throughout until 2 weeks after the last administration of study drug
6. Signed informed consent

Exclusion Criteria:

1. Decrease in size of the designated target ulcer(s) by ≥ 30% during the 7-day screening period
2. Cannot tolerate or comply with compression therapy.
3. An ulcer which shows signs of severe clinical infection, defined as pus oozing from the ulcer site
4. An ulcer positive for β-hemolytic streptococci upon culture
5. The ulcer has > 50% slough, significant necrotic tissue, bone, tendon, or capsule exposure or avascular ulcer beds
6. Is highly exuding (i.e. requires daily change of dressing)
7. Ankle brachial pressure index <0.65
8. Patients with active systemic infections
9. Patients with clinically significant medical conditions as determined by the investigator including renal, hepatic, hematologic, neurologic or immune disease. Examples include but are not limited to:

   1. Renal insufficiency as an estimated GFR which is < 30 mL/min/1.7m2
   2. Abnormal blood biochemistry defined as 3 times that of the upper limit of the normal range.
   3. Hepatic insufficiency defined as total bilirubin > 2 mg/dL or serum albumin < 25 g/L
   4. HbA1c > 9%
   5. Hemoglobin < 10 g/dL
   6. Hematocrit < 0.30
   7. Platelet count < 100,000
10. Presence of an active systemic or local cancer or tumor of any kind (with the exception of non-melanoma skin cancer)
11. Patients with severe rheumatoid arthritis (with more than 20 persistently inflamed joints, or below lower normal limit blood albumin level, or evidence of bone and cartilage damage on x-ray, or inflammation in tissues other than joints) and other collagen vascular diseases.
12. Patients with active connective tissue disease
13. Treatment with systemic corticosteroids (>15 mg/day), or current immunosuppressive agents
14. Previous or current radiation therapy or likelihood to receive this therapy during study participation
15. Pregnant or nursing patients
16. Known prior inability or unavailability to complete required study visits during study participation
17. Significant peripheral edema as per investigator's discretion
18. A psychiatric condition (e.g., suicidal ideation) or chronic alcohol or drug abuse problem, determined from the patient's medical history, which, in the opinion of the investigator, may pose a threat to patient compliance
19. Use of a platelet-derived growth factor within 28 days before screening
20. Use of any investigational drug or therapy within 28 days before screening
21. Has any other factor which may, in the opinion of the investigator, compromise participation and/or follow-up in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Measurement of aCT1 peptide (Active Pharmaceutical Ingredient in Granexin) levels in blood | Day 0
Measurement of aCT1 peptide (Active Pharmaceutical Ingredient in Granexin) levels in blood | Day 3
Measurement of aCT1 peptide (Active Pharmaceutical Ingredient in Granexin) levels in blood | Day 7

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Aiyan Diabetes Center, Augusta, Georgia
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Salem VA Medical Center, Salem, Virginia